CLINICAL TRIAL: NCT01924195
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Study of Anlotinib(AL3818) as Third Line Treatment in Patients With Advanced Non-small Cell Lung Cancer（ALTER0302）
Brief Title: Phase II Study of Anlotinib in Patients With Advanced Non-small Cell Lung Cancer（ALTER0302）
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALTN-03-II
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung; Anlotinib; AL3818; NSCLC; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anlotinib (Active Comparator): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo Capsule (Placebo Comparator): Placebo capsule QD po and it should be continued until disease progression or patients withdrawal of consent
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Anlotinib — Anlotinib QD po.
  Arms: Anlotinib
Drug: Placebo capsule — Placebo QD po.
  Arms: Placebo Capsule

SUMMARY:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit. It has the obvious resistance to new angiogenesis. The trial is to explore Anlotinib for the effectiveness and safety of andvanced non-small cell lung cancer who failed two lines of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. pathology diagnosed with advanced NSCL with measurable lesions;
2. Have failed for 2 lines of chemotherapy;
3. 18-70years,ECOG PS:0-2,Life expectancy of more than 3 months;
4. Other cytotoxic drugs,radiation therapy,or surgery≥4 weeks;
5. main organs function is normal;
6. must be agreed to take contraceptive measures during the study and within 6 months after end.

Exclusion Criteria:

1. SCLC(including mixed with NSCLC);
2. the central cavity of Squamous cell carcinoma and hemoptysis with NSCLC;
3. patients failed to use the anti-tumor angiogenesis therapy;
4. patients has many influence factors toward oral medications ;
5. Brain metastases patients accompanied by symptoms or symptom control for less than two months;
6. patients with severe and failed to controlled diseases,including: suboptimal blood pressure control;suffering from myocardial ischemia or above grade I myocardial infarction, arrhythmias and Class I heart failure;activity or failure to control severe infections;liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis;poorly controlled diabetes (FBG)>10mmol/L);urine protein≥++,etc.
7. patients failed to heal wounds or fractures for Long-term;
8. 4 weeks before enrollment, patients appeared NCI CTC AE grading >1 pulmonary hemorrhage; 4 weeks before enrollment, patients who appeared NCI CTC AE grade> 2 have other parts of the bleeding; patients has a tendency to bleed (eg active peptic ulcer) or are receiving thrombolytic or anticoagulant therapy such as warfarin, heparin or its analogues;
9. patients occurred venous thromboembolic events within 6 months;
10. patients has HIV-positive or organ transplantation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
enhanced CT/MRI scan | each 42 days up to disease progression
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT/MRI scan every two cycles. Refer to recist 1.1.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | each 21 days up to intolerance the toxicity(or PD)
  contain Serious Adverse Event To evaluate the safety of Anlotinib by CTC AE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Bao hui Han, doctor, Principal Investigator — Chest hospital affiliated to Shanghai jiaotong university
Locations (13):
- China (13):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing chest hospital，capital medical university, Beijing, Beijing Municipality
  - Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Jilin province tumor hospital, Changchun, Jilin
  - Shandong Province Tumor Hospital, Jinan, Shandong
  - Chest hospital affiliated to Shanghai jiaotong university, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The first affiliated hospital,zhejiang university, Hangzhou, Zhejiang